CLINICAL TRIAL: NCT02704039
Title: Multimodal Spectroscopy (MMS) for in Vivo Noninvasive Assessment of Skin
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Collaborators: Seton Healthcare Family (Other); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-07-0008
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this research program is to develop a simple, noninvasive diagnostic device for assessing skin pathology without the need for a biopsy. The device being studied is a single system capable of collecting three spectroscopy measurements (Raman, diffuse reflectance and laser induced fluorescence spectroscopy) from skin lesion sites. In order to accomplish this objective, the investigators propose to: 1) develop biophysical model for Raman spectroscopy of skin cancers, 2) conduct a clinical pilot study to collect MMS data from a minimum of 250 patients to determine the diagnostic accuracy (sensitivity and specificity) of MMS for diagnosing skin malignancy.

DETAILED DESCRIPTION:
To develop a biophysical model the investigators will recruit patients based on their known histopathology diagnoses, from each of 6 skin-cancer categories: basal cell carcinoma, squamous cell carcinoma, melanoma, atypical nevus, actinic keratosis, and benign skin. Patients with non-cancer diagnosis such as psoriasis, eczema / dermatitis, lichen planus or lupus will also be recruited. Recruitment will include 5 patients from each of these categories, giving a total of 20 patients. Measurements for the biophysical models are conducted on skin tissues that have been excised from the patients. Furthermore, these skin tissues are excised tissues that under standard screening procedure will be biopsied by the dermatologist. Therefore, patients are not undergoing extra & unnecessary biopsies, and will not be exposed to any risk involved with the microspectroscopy measurements.

To determine the diagnostic accuracy of MMS, MMS data will be collected from six clinical groups, each with a preoperative diagnosis: 1) malignant melanoma (MM), 2) basal cell carcinoma (BCC), 3) squamous cell carcinoma (SCC), 4) pre-cancerous lesions (AK), 5) benign or atypical nevi, or 6) other lesions or conditions (rare skin cancers such as merkel cell carcinoma, and inflammatory conditions such as psoriasis). The aim is to collect MMS data from a minimum of 240 patients (40 patients for each of the 6 groups), which will be split to training and validation datasets. Since several biopsies are required to diagnose a single skin cancer, it is anticipated that the actual number of pre-cancerous, benign and inflammatory lesions sampled will be much higher than our target total of 240, to be around 300. We will also collect data from non-skin cancer skin conditions: 1) psoriasis, 2) eczema / dermatitis, 3) lichen planus and 4) lupus. For the non-skin-cancer part of the study, we will enroll 20 patients from each of the categories, with a total target of 80 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing examination of skin
2. Male or Female 18 years and older
3. Patients with lesion(s) including one of the following: BCC, SCC, pre-cancerous, pigmented lesion, benign lesions, OR suspected diagnosis of psoriasis, eczema, dermatitis, lichen planus and/or lupus.
4. Signed consent form

Exclusion Criteria:

1. Patients with skin lesions in difficult to measure locations
2. Patients that do not sign the consent forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health adult volunteers being evaluated by dermatologist for lesion of interest (see inclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Aim 1: Develop biophysical model for Raman spectroscopy | 6 months
  use of a new technique of biophysical modeling to analyze the Raman spectra. At the core of the technique is the measurement of a set of "basis spectra" which are fit to the data using ordinary least-squares.
Aim 2: Perform clinical assessment of MMS for skin malignancy | 1 year
  develop a biophysically-orientated model of human skin using Raman spectroscopy, with the goal of obtaining tissue microenvironment structural and chemical information.

CONTACTS AND LOCATIONS:
Overall Officials: James Tunnell, PhD, Principal Investigator — University of Texas at Austin; Jason Reichenberg, MD, Principal Investigator — Seton & The University of Texas at Austin Dell Medical School
Locations (1):
- Seton Dermatology Clinics, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No